CLINICAL TRIAL: NCT00735566
Title: The Role of Endogenous Antiangiogenic Factors in Gastric Cancer Progression
Brief Title: Antiangiogenic Factors in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Jun Ho Lee, Staff Surgeon, National Cancer Center, Korea
Other Study IDs: NCCCTS 04-105
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; antiangiogenic factors; TNM stage
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for protein assay using ELISA
Oversight: Data Monitoring Committee: No

SUMMARY:
Endogenous antiangiogenic factors are related with gastric cancer progression.

DETAILED DESCRIPTION:
Gastric cancers have been known to secrete the proangiogenic cytokine VEGF in vitro and in vivo. Tumor VEGF expression is correlated with the severity of disease in patients with gastric cancer and some authors have suggested using circulating VEGF as a prognostic factor or tumor marker.In addition to producing proangiogenic cytokines, recent data demonstrate that tumors can produce antiangiogenic cytokine as well. It has been suggested that, in humans, the generation of antiangiogenic compounds in the presence of a primary tumor suppresses the growth of distant metastases. This phenomenon has been demonstrated in mice and in patients with clear cell renal cancer, breast cancer, and colorectal cancer. However, the presence of endogenous antiangiogenic cytokines in patients with gastric cancer has not been reported.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of gastric adenocarcinoma
* No other forms of cancer therapy, such as chemotherapy or radiotherapy for at least 3 weeks before the enrollment in study
* Performance status of 0, 1, 2 on the ECOG criteria
* ASA class I, II
* Patient compliance that allow adequate follow up
* Informed consent from patient or patient's relative.

Exclusion Criteria:

* Second primary malignancy
* EMR (Endoscopic mucosal resection) indication
* Laparoscopic gastrectomy
* Radiologic or clinical evidence of metastasis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible patients will undergo subtotal or total gastrectomy with D2 lymph node dissection
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Relationship between antiangiogenic factor and tumor, node, metastasis | One year

SECONDARY OUTCOMES:
Overall survival, treatment failure | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Lee, M.D., Ph.D, Principal Investigator — Gastric Cancer Branch, National Cancer Center
Locations (1):
- National Cancer Center, Goyang-si, Geonggi-do, South Korea